CLINICAL TRIAL: NCT05567445
Title: Characteristics and Outcomes of Heart Failure-Related Intensive Care Unit Admissions in Adults With Cardiomyopathy.
Brief Title: Outcome of Cardiomyopathic Adults Admission in ICU.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Abd-Elhmied Mohammed, Principal investigator, Assiut University
Other Study IDs: Cardiomyopathy in ICU.
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies | interventions — Echocardiography; Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples Without DNA — Blood for liver function, kideny function, CBC, BLOOD CULTURES.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography, CBC, Liver function, kideny function — Echocardiography, AST, ALT, UREA,CREAT. , CBC,may blood cultures.

SUMMARY:
To study the outcome of the cardiac function, and clinical status of the patiants with cardiomyopathy who are admitted in the I.C.U.

DETAILED DESCRIPTION:
Heart failure is not a single pathological diagnosis, but a clinical syndrome consisting of cardinal symptoms (e.g. breathlessness, ankle swelling, and fatigue) that may be accompanied by signs (e.g. elevated jugular venous pressure, pulmonary crackles, and peripheral oedema). It is due to a structural and/or functional abnormality of the heart that results in elevated intracardiac pressures and/or inadequate cardiac output at rest and/or during exercise. Identification of the aetiology of the underlying cardiac dysfunction is mandatory in the diagnosis of HF as the specific pathology can determine subsequent treatment. Most commonly, HF is due to myocardial dysfunction: either systolic, diastolic, or both. However, pathology of the valves, pericardium, and endocardium, and abnormalities of heart rhythm and conduction can also cause or contribute to HF.

Cardiomyopathies are defined by the WHO as diseases of the myocardium associated with cardiac dysfunction, Cardiomyopathies are categorized into dilated, restrictive, hypertrophic, and unclassified based on the predominant pathophysiologic characteristics. A new category has been added to include right ventricular abnormalities. The disorders that are associated with systemic or certain cardiac diseases are called specific heart muscle diseases and include ischemic cardiomyopathy, valvular, hypertensive, inflammatory, metabolic, peripartal, general systemic disease, muscular dystrophies, neuromuscular disorders, and toxic and hypersensitivity reactions. The unclassified cardiomyopathy category includes disorders such as fibroelastosis, noncompacted myocardium, and systolic dysfunction with minimal dilation.

Patiant admitted in I.C.U. with heart failure who already have cardiomyopathy Some patiants discharge without any comorbidies and some acquire renal failure, respiratory failure,MCS, sepsis, and some were associated with mortality . Significant comorbidities associated with these hospitalizations included arrhythmias, renal failure , cerebrovascular disease, and hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

Cardiomyopathic patiants admitted with heart failure diagonsed clinicaly , by Echocardiograph , or by ECG.

1. Dilated cardiomyopathy[ Unknown, Uremic cardiomyopathy, Post-partum, Ishemic].
2. Hypertrophic cardiomyopathy.
3. Acute heart failure caused by A.C.S. , Toxic myocardititis.

Exclusion Criteria:

1. Heart failure due to valvular heart disease.
2. Heart failure caused by hypertension.
3. patiant with COPD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiomyopathic patiants with the previous inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Effect on E.F. | through study completion, an average of 1 year
  Degree of impairement of E.F.
Effect on renal function | through study completion, an average of 1 year
  Who developed renal impairement, and its effect on cardiac function.
Sepsis | through study completion, an average of 1 year
  Who developed sepsis and its effect on cardiac function.
Effect on liver function | through study completion, an average of 1 year
  Who suffer liver function impairement, improvement or deteroriation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohammed Aly Obied-Allah, Ass.prof., Study Director — Assiut University; NoorEldeen Abd-El Azeem M.EL- Hefny, Prof, Study Director — Assiut University

REFERENCES:
- [Background] Seferovic PM, Polovina M, Bauersachs J, Arad M, Ben Gal T, Lund LH, Felix SB, Arbustini E, Caforio ALP, Farmakis D, Filippatos GS, Gialafos E, Kanjuh V, Krljanac G, Limongelli G, Linhart A, Lyon AR, Maksimovic R, Milicic D, Milinkovic I, Noutsias M, Oto A, Oto O, Pavlovic SU, Piepoli MF, Ristic AD, Rosano GMC, Seggewiss H, Asanin M, Seferovic JP, Ruschitzka F, Celutkiene J, Jaarsma T, Mueller C, Moura B, Hill L, Volterrani M, Lopatin Y, Metra M, Backs J, Mullens W, Chioncel O, de Boer RA, Anker S, Rapezzi C, Coats AJS, Tschope C. Heart failure in cardiomyopathies: a position paper from the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2019 May;21(5):553-576. doi: 10.1002/ejhf.1461. Epub 2019 Apr 16. PMID 30989768
- [Background] Rodriguez FH 3rd, Moodie DS, Parekh DR, Franklin WJ, Morales DL, Zafar F, Adams GJ, Friedman RA, Rossano JW. Outcomes of heart failure-related hospitalization in adults with congenital heart disease in the United States. Congenit Heart Dis. 2013 Nov-Dec;8(6):513-9. doi: 10.1111/chd.12019. Epub 2012 Nov 16. PMID 23164196
- [Background] Lange LG, Schreiner GF. Immune mechanisms of cardiac disease. N Engl J Med. 1994 Apr 21;330(16):1129-35. doi: 10.1056/NEJM199404213301607. PMID 8133856
- [Background] Matsubara I, Tedo I. [Study on the respiratory failure with cardiac failure--focus on hypoventilation respiratory failure]. Kokyu To Junkan. 1990 Aug;38(8):785-9. Japanese. PMID 2218087
- [Background] Platz E, Jhund PS, Claggett BL, Pfeffer MA, Swedberg K, Granger CB, Yusuf S, Solomon SD, McMurray JJ. Prevalence and prognostic importance of precipitating factors leading to heart failure hospitalization: recurrent hospitalizations and mortality. Eur J Heart Fail. 2018 Feb;20(2):295-303. doi: 10.1002/ejhf.901. Epub 2017 Sep 4. PMID 28872259
- [Background] Ahmed A, Allman RM, Fonarow GC, Love TE, Zannad F, Dell'italia LJ, White M, Gheorghiade M. Incident heart failure hospitalization and subsequent mortality in chronic heart failure: a propensity-matched study. J Card Fail. 2008 Apr;14(3):211-8. doi: 10.1016/j.cardfail.2007.12.001. PMID 18381184
- [Background] van Deursen VM, Damman K, Hillege HL, van Beek AP, van Veldhuisen DJ, Voors AA. Abnormal liver function in relation to hemodynamic profile in heart failure patients. J Card Fail. 2010 Jan;16(1):84-90. doi: 10.1016/j.cardfail.2009.08.002. Epub 2009 Sep 26. PMID 20123323
- See also: Heart failure and sepsis: practical recommendations for the optimal management — https://link.springer.com/article/10.1007/s10741-019-09816-y
- See also: Heart Failure in Acute Ischemic Stroke — https://www.ingentaconnect.com/content/ben/ccr/2010/00000006/00000003/art00008